CLINICAL TRIAL: NCT01384708
Title: Evaluation of a Miniaturized Microscope Device for the Detection of Esophageal Squamous Cell Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anandasabapathy, Sharmila, M.D. (Individual)
Collaborators: William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GCO# 10-0982
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2014-03

CONDITIONS: Squamous Cell Cancer
Keywords: squamous cell cancer; squamous cell neoplasia
MeSH Terms: conditions — Neoplasms, Squamous Cell | interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): imaging with proflavine
  Interventions: Drug: proflavine

INTERVENTIONS:
Drug: proflavine — 1-10 ml of proflavine (derived form dissolving 10mg proflavine hemisulfate USP in 100 ml sterile water)
  Other Names: Proflavine hemisulfate

SUMMARY:
The overall objective of this study is to determine whether high-resolution imaging of the esophagus during routine diagnostic upper endoscopy can assist clinicians in detecting and discriminating dysplastic (precancerous) areas. This high-resolution microendoscope (HRME) was developed by our collaborators at Rice University and provides > 1000x magnified images of the esophageal mucosa. The purpose of this study is to determine whether this device can be used to enhance the diagnostic accuracy of routine endoscopic screening for squamous cell cancer of the esophagus.

ELIGIBILITY:
Inclusion Criteria:

* known or suspected squamous cell neoplasia
* 18 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
to determine whether or not tissue is neoplastic or non-neoplastic | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Protano MA, Xu H, Wang G, Polydorides AD, Dawsey SM, Cui J, Xue L, Zhang F, Quang T, Pierce MC, Shin D, Schwarz RA, Bhutani MS, Lee M, Parikh N, Hur C, Xu W, Moshier E, Godbold J, Mitcham J, Hudson C, Richards-Kortum RR, Anandasabapathy S. Low-Cost High-Resolution Microendoscopy for the Detection of Esophageal Squamous Cell Neoplasia: An International Trial. Gastroenterology. 2015 Aug;149(2):321-329. doi: 10.1053/j.gastro.2015.04.055. Epub 2015 May 14. PMID 25980753